CLINICAL TRIAL: NCT03960567
Title: Evaluation of the Accuracy and the Intra and Inter Rater Reliability of the POGO Score
Brief Title: Evaluation of the Accuracy of the POGO Score
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Assoc Prof, Diskapi Teaching and Research Hospital
Other Study IDs: POGO
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-05

CONDITIONS: Intubation
Keywords: Intubation; Laryngeal view; Scoring systems; Larynx
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Videolaryngoscopy — Patient will be intubated by using videolaryngoscope

SUMMARY:
A classification method describing the larynx appearance during laryngoscopy accepted by all anesthetists has not been defined yet. In one study, it was shown that anesthetists mis classed the glottis image by 50%. The most commonly used classification method is the Cormack Lehane (CL) classification. This classification classifies the larynx appearance during direct laryngoscopy form 1 to 4. The modified CL classification is criticized as it does not predict difficult intubation and especially grade 2 is operator dependent and partial view is not well defined. The numerical expression of the percentage of the glottic aperture (POGO = percentile of glottic opening) is another score. In this score, A POGO score of 100% accounts for full visualization of the larynx starting from anterior commissure to the posterior cartilage, while 0% indicated a complete absence of glottic opening.

The use of a standard and effective classification method will facilitate and accelerate communication between anesthetists in difficult life-threatening situations such as difficult airway / difficult intubation / difficult ventilation and contribute to patient safety. The use of common terminology can also facilitate the evaluation of the performance of intubation tools.

The aim of this study was to evaluate the accuracy and intra and inter rater reliability of the POGO score.

DETAILED DESCRIPTION:
Anesthesiologist will be asked to score still images of laryngeal views, which will be obtained from patients requiring intubation for general anesthesia, after obtaining written informed consent.

The images of the larynx will be captured first with the Macintosh blade and thereafter with the D blade. A group of independent anesthesiologist will score these images with the Cormack Lehane and POGO scores. The set of images will be prepared from patients with both difficult and normal airway anatomy. Some images in the series will be repeated to assess intra rater variability.

The anesthesiologist will be asked to rate 20 images both with the CL and POGO scores.

The experience of the raters in airway management, their experience with videolaryngoscopy and scoring systems used currently when documenting videolaryngoscopy and demographic data will be also obtained.

The POGO scores of the participants and investigators will be compared.

The outcome of interest is the correct POGO score rate of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving general anesthesia

Exclusion Criteria:

* Emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery and those who are intubated
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Percentile of glottic opening | 2 minutes after induction of anesthesia
  A percentile of glottic opening score of 100% accounts for full visualization of the larynx starting from anterior commissure to the posterior cartilage, while 0% indicated a complete absence of glottic opening.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ünal, Assoc. Prof., Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- Dilek Ünal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yentis SM, Lee DJ. Evaluation of an improved scoring system for the grading of direct laryngoscopy. Anaesthesia. 1998 Nov;53(11):1041-4. doi: 10.1046/j.1365-2044.1998.00605.x. PMID 10023271
- [Background] Norris A, Heidegger T. Limitations of videolaryngoscopy. Br J Anaesth. 2016 Aug;117(2):148-50. doi: 10.1093/bja/aew122. Epub 2016 Jun 1. No abstract available. PMID 27251753
- [Background] Ochroch EA, Hollander JE, Kush S, Shofer FS, Levitan RM. Assessment of laryngeal view: percentage of glottic opening score vs Cormack and Lehane grading. Can J Anaesth. 1999 Oct;46(10):987-90. doi: 10.1007/BF03013137. PMID 10522589
- [Background] Roznovan VK. [Condition of oxidation-reduction processes in patients with chronic osteomyelitis of the jaw and phlegmons of the maxillofacial area in connection with surgical intervention and anesthesia]. Stomatologiia (Mosk). 1975 Jan-Feb;54(1):33-6. No abstract available. Russian. PMID 1054169
- [Background] Cook TM. A grading system for direct laryngoscopy. Anaesthesia. 1999 May;54(5):496-7. doi: 10.1046/j.1365-2044.1999.0907f.x. No abstract available. PMID 10995154